CLINICAL TRIAL: NCT07406763
Title: Effect of Adding Blood Flow Restriction to Traditional Program After Anterior Cruciate Ligament Reconstruction: A Double-Blinded Randomized Controlled Trial
Brief Title: Blood Flow Restriction in ACL Reconstruction Rehabilitation: A Double-Blinded RCT
Acronym: *BFR*
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Mohamed Mahmoud Abdelaziz Khalil (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Ahmed Mohamed Mahmoud Abdelaziz Khalil, doctor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003141
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Blood Flow Restriction Therapy; Anterior Cruciate Ligament (ACL)
Keywords: ACLR; BFRT
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: patient and research assistant (the examiner of all patients) were blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Rehabilitation Protocol Group (Active Comparator): Participants in this group received a standard postoperative rehabilitation program following anterior cruciate ligament reconstruction (ACLR) from the 2nd to the 12th postoperative week.
  Interventions: Other: traditional rehabilitation protocol
- Blood Flow Restriction (BFR) plus Traditional Rehabilitation Group (Experimental): Participants in this group received the same traditional postoperative rehabilitation protocol as the control group from the 2nd to the 12th postoperative week, with the addition of blood flow restriction (BFR) training applied during selected strengthening exercises.
  Interventions: Other: traditional rehabilitation protocol; Device: Blood Flow Restriction

INTERVENTIONS:
Other: traditional rehabilitation protocol — The traditional rehabilitation protocol includes progressive therapeutic exercises aimed at restoring:
  Quadriceps and hamstring muscle strength Knee joint range of motion Neuromuscular control and functional performance
Device: Blood Flow Restriction — Blood flow restriction was applied to the proximal thigh of the operated limb using a specially designed sphygmomanometer cuff capable of partially restricting arterial inflow and venous outflow during exercise. BFR was used during low-load resistance exercises targeting the quadriceps and hamstring muscles, in accordance with postoperative safety guidelines.
  Arms: Blood Flow Restriction (BFR) plus Traditional Rehabilitation Group

SUMMARY:
The goal of this clinical trial is to learn whether adding blood flow restriction (BFR) training to a traditional rehabilitation protocol (TRP) can improve muscle strength, knee proprioception, range of motion, pain, and lower limb function after anterior cruciate ligament reconstruction (ACLR).

This study is conducted in male and female adults aged 18-35 years who underwent ACLR using a semitendinosus tendon autograft.

The main questions it aims to answer are:

Does adding BFR to a traditional rehabilitation protocol improve quadriceps and hamstring muscle strength after ACLR? Does adding BFR improve knee joint proprioception, range of motion, pain, and lower limb function after ACLR? Researchers compared a traditional rehabilitation protocol alone (control group) with the same protocol combined with blood flow restriction training (BFR group) to see if BFR provides superior improvements in postoperative outcomes.

Participants was: randomly assigned to either a traditional rehabilitation group or a BFR-assisted rehabilitation group Perform supervised rehabilitation exercises from the 2nd to the 12th postoperative week Undergo assessments of muscle strength, knee proprioception, range of motion, pain, and function Be evaluated 1 week before surgery and at 1.5 and 3 months after ACL reconstruction

DETAILED DESCRIPTION:
Anterior cruciate ligament reconstruction (ACLR) is commonly followed by persistent quadriceps and hamstring weakness, reduced knee range of motion, impaired proprioception, pain, and limitations in lower limb function despite standard rehabilitation. Traditional postoperative rehabilitation protocols may not fully restore neuromuscular performance within the early months following surgery.

Blood flow restriction (BFR) training has emerged as a rehabilitation strategy that allows low-load exercise to produce strength gains comparable to high-load training by partially restricting arterial inflow and venous outflow during exercise. This approach may be particularly beneficial in the early postoperative phase after ACLR, when high mechanical loading is contraindicated.

This randomized controlled clinical trial investigates the effects of adding BFR training to a traditional rehabilitation protocol following ACL reconstruction. Participants are randomly allocated to either a traditional rehabilitation protocol alone or the same protocol combined with BFR applied to the operated limb during exercise sessions. Rehabilitation is initiated in the early postoperative period and continues for a standardized duration.

Clinical outcomes related to muscle performance, knee joint function, proprioceptive accuracy, range of motion, and pain are evaluated at multiple time points before and after surgery to examine short-term and mid-term recovery patterns. The study aims to determine whether the inclusion of BFR enhances functional recovery compared with conventional rehabilitation alone following ACLR.

ELIGIBILITY:
Inclusion Criteria Male or female participants aged 18-35 years Undergoing primary unilateral anterior cruciate ligament reconstruction Reconstruction performed using semitendinosus tendon autograft Referred for postoperative rehabilitation by an orthopedic surgeon Medically cleared to participate in postoperative rehabilitation and exercise training Ability to understand and follow verbal instructions Willingness to participate and provide written informed consent Exclusion Criteria History of previous surgery on either knee Concomitant ligament injuries requiring surgical repair (e.g., PCL, MCL, LCL) Severe meniscal injury requiring repair or affecting rehabilitation progression Known cardiovascular, vascular, or thromboembolic disorders Peripheral vascular disease or conditions contraindicating blood flow restriction training Neurological disorders affecting lower limb function Uncontrolled systemic disease (e.g., uncontrolled diabetes or hypertension) Postoperative complications such as infection, deep vein thrombosis, or graft failure Inability to comply with the rehabilitation program or follow-up assessments

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Quadriceps Muscle Strength | preoperative baseline, 1.5 months post-operative, and 3 months post-operative
  Assessed using a handheld dynamometer (HHD) Measured on the operated limb
Hamstring Muscle Strength | preoperative baseline, 1.5 months post-operative, and 3 months post-operative
  Assessed using a handheld dynamometer (HHD) Measured on the operated limb

SECONDARY OUTCOMES:
Knee Joint Proprioception (Joint Position Sense) | preoperative baseline, 1.5 months post-operative, and 3 months post-operative
  Assessed using a digital inclinometer Evaluated as joint position sense accuracy
Knee Joint Range of Motion (ROM) | preoperative baseline, 1.5 months post-operative, and 3 months post-operative
  Flexion and extension measured using a digital goniometer
Knee Joint Pain | preoperative baseline, 1.5 months post-operative, and 3 months post-operative
  Assessed using the Visual Analog Scale (VAS)
Lower Limb Function | preoperative baseline, 1.5 months post-operative, and 3 months post-operative
  Assessed using the Arabic version of the Lower Extremity Functional Scale (LEFS)

CONTACTS AND LOCATIONS:
Overall Officials: Maha Mohammed, A.Prof, Study Director — Cairo University
Locations (2):
- Egypt (2):
  - Cairo University, Cairo, Cairo Governorate
  - Physical Therapy, Giza

IPD SHARING:
Plan to Share IPD: No
Not applicable - the thesis does not describe a plan to share individual participant data with other researchers.

REFERENCES:
- [Result] Abe T, Kearns CF, Sato Y. Muscle size and strength are increased following walk training with restricted venous blood flow from the leg muscle, Kaatsu-walk training. J Appl Physiol (1985). 2006 May;100(5):1460-6. doi: 10.1152/japplphysiol.01267.2005. Epub 2005 Dec 8. PMID 16339340
- [Result] Kramer LC, Denegar CR, Buckley WE, Hertel J. Factors associated with anterior cruciate ligament injury: history in female athletes. J Sports Med Phys Fitness. 2007 Dec;47(4):446-54. PMID 18091686
- [Result] Elwood PC, Pickering J, Bayer A, Gallacher JE. Vascular disease and cognitive function in older men in the Caerphilly cohort. Age Ageing. 2002 Jan;31(1):43-8. doi: 10.1093/ageing/31.1.43. PMID 11850307
- [Result] Yip T, Wang Y, Mootoo C, Mirpuri S. Moderating the association between discrimination and adjustment: A meta-analysis of ethnic/racial identity. Dev Psychol. 2019 Jun;55(6):1274-1298. doi: 10.1037/dev0000708. Epub 2019 Mar 25. PMID 30907605
- [Result] Pletch A, Morcuende J, Barriga H, Segura J, Salas A. Photovoice and Clubfoot: Using a Participatory Research Method to Study Caregiver Adherence to the Ponseti Method in Peru. Iowa Orthop J. 2015;35:160-8. PMID 26361460
- [Result] Lepley AS, Grooms DR, Burland JP, Davi SM, Kinsella-Shaw JM, Lepley LK. Quadriceps muscle function following anterior cruciate ligament reconstruction: systemic differences in neural and morphological characteristics. Exp Brain Res. 2019 May;237(5):1267-1278. doi: 10.1007/s00221-019-05499-x. Epub 2019 Mar 9. PMID 30852644
- [Result] Herring AA, Stone MB, Frenkel O, Chipman A, Nagdev AD. The ultrasound-guided superficial cervical plexus block for anesthesia and analgesia in emergency care settings. Am J Emerg Med. 2012 Sep;30(7):1263-7. doi: 10.1016/j.ajem.2011.06.023. Epub 2011 Oct 24. PMID 22030184
- [Result] Laurentino GC, Loenneke JP, Mouser JG, Buckner SL, Counts BR, Dankel SJ, Jessee MB, Mattocks KT, Iared W, Tavares LD, Teixeira EL, Tricoli V. Validity of the Handheld Doppler to Determine Lower-Limb Blood Flow Restriction Pressure for Exercise Protocols. J Strength Cond Res. 2020 Sep;34(9):2693-2696. doi: 10.1519/JSC.0000000000002665. PMID 29912080
- [Result] Schlag J, Pouget A, Sadeghpour S, Schlag-Rey M. Interactions between natural and electrically evoked saccades. III. Is the nonstationarity the result of an integrator not instantaneously reset? J Neurophysiol. 1998 Feb;79(2):903-10. doi: 10.1152/jn.1998.79.2.903. PMID 9463451
- [Result] Felszeghy S, Modis L, Nemeth P, Nagy G, Zelles T, Agre P, Laurikkala J, Fejerskov O, Thesleff I, Nielsen S. Expression of aquaporin isoforms during human and mouse tooth development. Arch Oral Biol. 2004 Apr;49(4):247-57. doi: 10.1016/j.archoralbio.2003.09.011. PMID 15003543
- [Result] Krych AJ, Pitts RT, Dajani KA, Stuart MJ, Levy BA, Dahm DL. Surgical repair of meniscal tears with concomitant anterior cruciate ligament reconstruction in patients 18 years and younger. Am J Sports Med. 2010 May;38(5):976-82. doi: 10.1177/0363546509354055. Epub 2010 Mar 18. PMID 20299545
- [Result] Liu A, Xue GH, Sun M, Shao HF, Ma CY, Gao Q, Gou ZR, Yan SG, Liu YM, He Y. 3D Printing Surgical Implants at the clinic: A Experimental Study on Anterior Cruciate Ligament Reconstruction. Sci Rep. 2016 Feb 15;6:21704. doi: 10.1038/srep21704. PMID 26875826
- [Result] Lindstrom M, Strandberg S, Wredmark T, Fellander-Tsai L, Henriksson M. Functional and muscle morphometric effects of ACL reconstruction. A prospective CT study with 1 year follow-up. Scand J Med Sci Sports. 2013 Aug;23(4):431-42. doi: 10.1111/j.1600-0838.2011.01417.x. Epub 2011 Nov 23. PMID 22107159
- [Result] Loenneke JP, Abe T, Wilson JM, Thiebaud RS, Fahs CA, Rossow LM, Bemben MG. Blood flow restriction: an evidence based progressive model (Review). Acta Physiol Hung. 2012 Sep;99(3):235-50. doi: 10.1556/APhysiol.99.2012.3.1. PMID 22982712
- [Result] Malinzak RA, Colby SM, Kirkendall DT, Yu B, Garrett WE. A comparison of knee joint motion patterns between men and women in selected athletic tasks. Clin Biomech (Bristol). 2001 Jun;16(5):438-45. doi: 10.1016/s0268-0033(01)00019-5. PMID 11390052
- [Result] Marcon M, Ciritsis B, Laux C, Nanz D, Nguyen-Kim TD, Fischer MA, Andreisek G, Ulbrich EJ. Cross-sectional area measurements versus volumetric assessment of the quadriceps femoris muscle in patients with anterior cruciate ligament reconstructions. Eur Radiol. 2015 Feb;25(2):290-8. doi: 10.1007/s00330-014-3424-2. Epub 2014 Oct 31. PMID 25358592
- [Result] May AK, Brandner CR, Warmington SA. Hemodynamic responses are reduced with aerobic compared with resistance blood flow restriction exercise. Physiol Rep. 2017 Feb;5(3):e13142. doi: 10.14814/phy2.13142. PMID 28183863
- [Result] McHugh MP, Tyler TF, Gleim GW, Nicholas SJ. Preoperative indicators of motion loss and weakness following anterior cruciate ligament reconstruction. J Orthop Sports Phys Ther. 1998 Jun;27(6):407-11. doi: 10.2519/jospt.1998.27.6.407. PMID 9617726
- [Result] Minniti MC, Statkevich AP, Kelly RL, Rigsby VP, Exline MM, Rhon DI, Clewley D. The Safety of Blood Flow Restriction Training as a Therapeutic Intervention for Patients With Musculoskeletal Disorders: A Systematic Review. Am J Sports Med. 2020 Jun;48(7):1773-1785. doi: 10.1177/0363546519882652. Epub 2019 Nov 11. PMID 31710505
- [Result] Ozaki H, Sakamaki M, Yasuda T, Fujita S, Ogasawara R, Sugaya M, Nakajima T, Abe T. Increases in thigh muscle volume and strength by walk training with leg blood flow reduction in older participants. J Gerontol A Biol Sci Med Sci. 2011 Mar;66(3):257-63. doi: 10.1093/gerona/glq182. Epub 2010 Oct 25. PMID 20974731
- [Result] Relph N, Herrington L, Tyson S. The effects of ACL injury on knee proprioception: a meta-analysis. Physiotherapy. 2014 Sep;100(3):187-95. doi: 10.1016/j.physio.2013.11.002. Epub 2013 Dec 4. PMID 24690442
- [Result] Zou W, Cheng H, Li S, Yue X, Xue Y, Chen S, Kang L. Polymodal Responses in C. elegans Phasmid Neurons Rely on Multiple Intracellular and Intercellular Signaling Pathways. Sci Rep. 2017 Feb 14;7:42295. doi: 10.1038/srep42295. PMID 28195191
- [Result] van der Made AD, Paget LDA, Altink JN, Reurink G, Six WR, Tol JL, Kerkhoffs GM. Assessment of Isometric Knee Flexor Strength Using Hand-Held Dynamometry in High-Level Rugby Players Is Intertester Reliable. Clin J Sport Med. 2021 Sep 1;31(5):e271-e276. doi: 10.1097/JSM.0000000000000793. PMID 31842051
- [Result] Suga T, Okita K, Takada S, Omokawa M, Kadoguchi T, Yokota T, Hirabayashi K, Takahashi M, Morita N, Horiuchi M, Kinugawa S, Tsutsui H. Effect of multiple set on intramuscular metabolic stress during low-intensity resistance exercise with blood flow restriction. Eur J Appl Physiol. 2012 Nov;112(11):3915-20. doi: 10.1007/s00421-012-2377-x. Epub 2012 Mar 14. PMID 22415101
- [Result] Abe T, Fujita S, Nakajima T, Sakamaki M, Ozaki H, Ogasawara R, Sugaya M, Kudo M, Kurano M, Yasuda T, Sato Y, Ohshima H, Mukai C, Ishii N. Effects of Low-Intensity Cycle Training with Restricted Leg Blood Flow on Thigh Muscle Volume and VO2MAX in Young Men. J Sports Sci Med. 2010 Sep 1;9(3):452-8. eCollection 2010. PMID 24149640
- See also: After inclusion in the study, every patient signed an informed consent form , and then was randomly assigned to one of the two groups using a random generator — https://www.random.org